CLINICAL TRIAL: NCT03380312
Title: Prospective Cohort Study on Mesh Shrinkage Measured with MRI After Robot Assisted Laparoscopic Retromuscular Hernia Repair Using an Iron Oxide Loaded PVDF Mesh
Brief Title: MRI Imaging of Ipsilateral Retromuscular Access
Status: Completed | Type: Observational
Sponsor: Filip Muysoms (Other)
Responsible Party: Sponsor-Investigator, Filip Muysoms, Surgeon, Algemeen Ziekenhuis Maria Middelares
Organization: Algemeen Ziekenhuis Maria Middelares (Other)
Other Study IDs: IRMA
Record Dates: First submitted 2017-12-06; First posted 2017-12-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-03

CONDITIONS: Hernia, Incisional
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: rTARUP technique — robot-assisted rTARUP technique

SUMMARY:
The aim of this study is to measure the mesh shrinkage and the visualization of the mesh with MRI scan at 1 month and 13 months after robot assisted retromuscular incisional hernia repair with ipsilateral access and the use of the visible CICAT mesh (Dynamesh®) for defect repair. The investigators also want to measure the volume of the rectus muscles and the change between 1 and 13 months.

DETAILED DESCRIPTION:
The aim of this study is to measure the mesh shrinkage and the visualization of the mesh with MRI scan at 1 month and 13 months after robot assisted retromuscular incisional hernia repair with ipsilateral access and the use of the visible CICAT mesh (Dynamesh®) for defect repair. The investigators also want to measure the volume of the rectus muscles and the change between 1 and 13 months. Possibly the ipsilateral retromuscular access could induce some atrophy of the rectus muscles.

The study will be conducted in the department of surgery in het AZ Maria Middelares, Ghent, Belgium. Dr. Filip Muysoms will personally select and operate all patients eligible for this study. Dr.Muysoms will inform all patients about the surgery and the follow-up with MRI scan thereafter. Dr. Beckers and Dr. Heindryckx will perform all MRI examinations of the patients at 1 month and 13 months post-operatively and will be available for questions from the patient.

The investigators want to show that with this type of mesh it is possible to visualize the mesh after retromusculare placement in vivo in a safe manner. Furthermore, the positioning of the mesh, mesh shrinkage or mesh shifting will be monitored with this technique. This provides long-term benefit and provides early treatment possibilities in case of post-operative complications related to the mesh position.

ELIGIBILITY:
Inclusion Criteria:

* 20 patients selected and operated by PI.

Exclusion Criteria:

* <18 years
* Emergency surgery (incarcerated hernia)
* Clean-contaminated, contaminated or dirty procedures (according to the CDC classification)
* Lateral hernias
* Hernias that need a component separation technique.
* Previous mesh repair on the midline
* ASA score> 4
* Pregnancy
* No patient Informed Consent
* Life expectancy of less than 2years
* Contraindications for MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients scheduled for robot assisted laparoscopic retromuscular repair (rTARUP =robotic Trans Abdominal Retromuscular Umbilical Prosthesis) of a midline ventral hernia will be invited to take part in the study. Both primary ventral and incisional midline hernias will be included (EHS classification M1-M5).
  A total of 20 patients will be enrolled in this observational study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2021-06-19 (Actual); Study Completion 2022-01-19 (Actual)

PRIMARY OUTCOMES:
Change of the mesh surface (percentage) | 1 month and 13 month post-operatively
  Shrinkage rate / change of the mesh surface (percentage) as measured with the MRI between 1 month and 13 months postoperatively, defined as (100 - mesh surface at 13 months x 100 / mesh surface at 1 month)

SECONDARY OUTCOMES:
Change in mesh surface between implantation surface size | 1 month and 13 month post-operatively
  Change in mesh surface between implantation surface size, surface at 1m and at 13m
Change in mesh width and length between implantation surface size | 1 month and 13 month post-operatively
  Change in mesh width and length between implantation surface size, surface at 1m and at 13m
Volume of the rectus muscle at the level of the umbilicus | 1 month and 13 month post-operatively
  Volume of the rectus muscle at the level of the umbilicus on both sides at 1m and at 13m
Operation duration | once during operation
  recording of the operation duration needed for robo-assisted TARUP
Intra-operative complications | until 4 weeks post-operative
  Intra-operative complications registered until 4 weeks after the hernia repair
Early post-operative complications | until 30 days post-operative
  Early post-operative complications detected until 30 days after hernia repair
Late complications | after 30 days post-operative
  Late complications (after 30 days)
Quality of Life questionnaire | preoperative and 1 month and 13 month post-operatively
  A questionnaire will be used to measured life quality of the participants preoperatively and at 1m and 13m postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Filip Muysoms, MD,PhD, Principal Investigator — Algemeen Ziekenhuis Maria Middelares
Locations (1):
- AZ Maria Middelares, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vierstraete M, Beckers R, Vangeel L, Foriers B, Pletinckx P, Muysoms F. Prospective cohort study on mesh shrinkage measured with MRI after robot-assisted minimal invasive retrorectus ventral hernia repair using an iron-oxide-loaded polyvinylidene fluoride mesh. Surg Endosc. 2023 Jun;37(6):4604-4612. doi: 10.1007/s00464-023-09938-3. Epub 2023 Feb 28. PMID 36854798